CLINICAL TRIAL: NCT03660722
Title: Bone, Inflammation, Gut and Renal Biomarkers in Antiretroviral Naïve HIV-1 Positive Subjects Commencing Antiretroviral Therapy: the BIGgeR Study.
Brief Title: Bone, Inflammation, Gut and Renal Biomarkers in Antiretroviral Naïve HIV-1 Positive Subjects
Acronym: BIGGER
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study not started
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1708212; 2018-001358-84 (EudraCT Number)
Record Dates: First submitted 2018-09-04; First posted 2018-09-06 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: HIV Positive
MeSH Terms: conditions — HIV Seropositivity | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Blood and urinary sample (Other): Blood and urinary sample in HIV 1 positive adults initiating treatment
  Interventions: Other: blood and urinary samples

INTERVENTIONS:
Other: blood and urinary samples — blood samples, rectal and urethral swabs , urine samples at inclusion, after 4 weeks then 12 weeks

SUMMARY:
Co-morbidities, including low bone mineral density, increased visceral adiposity and chronic kidney disease (CKD) are frequent in people living with HIV, and may be driven by ongoing inflammation and immune activation. Initiation of ART reduces inflammation and immune activation and is associated with changes in bone and renal biomarkers and gut microbiota. Investigators hypothesise that changes in gut microbiome when starting antiretroviral therapy correlate to changes in bone and renal biomarkers and wish to explore possible mechanisms linking these by investigating changes in markers of inflammation and immune activation.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 positive
* Age 18-64 years
* Able to give informed consent
* Not previously treated for chronic HIV-1 infection, except for pre- or post- exposure prophylaxis exposure or treatment for mother to child transmission >12 months ago
* Due to commence antiretroviral therapy by treating clinician

Exclusion Criteria:

* - Previous major intestinal surgery/inflammatory bowel conditions
* Infective diarrhoea in the last 3 months
* BMI<18.5
* Currently pregnant OR planning to conceive during the study period
* Previous use of antiretroviral therapy, except for pre- or post- exposure prophylaxis exposure or treatment for mother to child transmission >12 months ago
* Use of antibiotics (except for prophylactic co-trimoxazole) within the last 2 months

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
faecal microbial alpha-diversity | At 12 weeks
  Change in faecal microbial alpha-diversity (change in mean Shannon Diversity Index score in faecal microbiota) .

SECONDARY OUTCOMES:
markers of gut epithelium integrity | At 12 weeks
  Change in markers of gut epithelium integrity and bacterial translocation
inflammatory marker | at 12 weeks
  Change in inflammatory marker (c-reactive protein)
circulating markers of monocyte activation | at 12 weeks
  Change in circulating marker of monocyte activation
renal glomerular biomarkers | at 12 weeks
  Change in renal glomerular biomarker (KIM-1)
bone biomarkers | at 12 weeks
  Change in bone biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Amandine GAGNEUX-BRUNON, MD, Principal Investigator — CHU SAINT-ETIENNE
Locations (1):
- Chu Saint-Etienne, Saint-Etienne, France

IPD SHARING:
Plan to Share IPD: No